CLINICAL TRIAL: NCT01356589
Title: Retrospective Study on Intrapatient VAriabiLity of the Hemoglobin Levels in Anemic CKD Patients in Predialysis (Stage 3-4) and Dialysis (Stage 5) Treated With MIRCERA® (RIVAL Study)
Brief Title: A Study of MIRCERA for the Intrapetient Variability of Hemoglobin Levels in Patients With Chronic Renal Anemia (RIVAL)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25289
Record Dates: First submitted 2011-05-18; First posted 2011-05-19 (Estimated); Results first posted 2015-12-28 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This retrospective observational study will assess the incidence of hemoglobin cycling in chronic kidney disease (stage 3, 4, and 5) patients with renal anemia treated with Mircera (methoxy polyethylene glycol-epoetin beta). Data will be collected from each patient from a 9-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic kidney disease in predialysis (stage 3 and 4) and dialysis
* Renal anemia treated with Mircera according to label for at least 9 months before date of signed informed consent

Exclusion Criteria:

* Participation in an interventional clinical trial within the retrospective observation period
* Contraindications to Mircera administration as per label or judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease patients with anemia treated with Mircera
Sampling Method: Probability Sample
Enrollment: 1288 (Actual)
Dates: Start 2010-09-30 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- Greece (33):
  - Timios Stavros Clinic; Nephrology Department, Aigáleo
  - General Hospital of Artas; Nephrology, Arta
  - Attikon Center; Nephrology, Athens
  - Athinaiki Private Clinic, Athens
  - Hospital henry dunant; Nephrology, Athens
  - General Hospital Hippokration of Athens; Nephrology, Athens
  - General Hospital Of Athens G.Gennimatas; Nephrology, Athens
  - Kyanos Stavros Private Hospital; Nephrologic Clinic, Athens
  - General Hospital Of West Attikis; Nephrology, Athens
  - University Hospital Attikon ; Pathology Clinic, Athens
  - General Hospital Agia Olga; Nephrology, Athens
  - Iaso General Private Clinic; Nephrology, Athens
  - Iatriko Athinon Clinic Dafnis; Nephrology Department, Daphni-athens
  - General Hospital Of Dramas; Dialysis Center Unit, Drama
  - University Hospital Of Heraklion; Nefrologiki Clinic, Heraklion
  - General Hospital Of Katerinis; Nephrology Unit, Katerini
  - General Hospital Of Lamias; Nephrology, Lamia
  - Univeristy Hospital of Larissa; Nephrology, Larissa
  - Eytychios Patsidis Center Of Haemodialysis, Larissa
  - General Hospital Of Leykadas; Dialysis Center Unit, Leykada
  - Leivadia General Hospital; Nephrologic Clinic, Livadeia
  - Kyanous Stavros of Patras, Renal Disease Therapy Unit, Pátrai
  - Olympion Therapeytirion; Nefrology, Pátrai
  - General Hospital Tzanio ; Nephrology, Piraeus
  - General Hospital Of Chalkidikis; Dialysis Center Unit, Polygyros
  - Rodos General Hospital; Nephrologic Clinic, Rhodes
  - Alpha Nephrodynamiki Of Serres; Dialysis Center Unit, Serres
  - Ahepa Hospital; 1St Dept. of Medicine, Thessaloniki
  - IPPOKRATES Private Dialysis Centre, Thessaloniki
  - General Hospital Of Thessalonikis Papageorgiou; Nephrology, Thessaloniki
  - Alfa Nefrodynamiki; Nefrology, Thessaloniki
  - Thessaliki Nossileytiki; Nephrology, Volos
  - General Hospital of Volos; Nephrology, Volos

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera: Participants with renal anemia due to chronic kidney disease (CKD) in pre-dialysis (Stage 3-4) and dialysis (Stage 5) were treated with Mircera according to the label for at least 9 months. This non-interventional study did not affect by any means the treatment, medical care or monitoring of the participant, since it reported 9-month retrospective data, which already existed in the participants' medical files.
Period: Overall Study
Arm/Group | Mircera
Started | 1288
Treated | 1285
Completed | 1283
Not Completed | 5
Not completed — Enrolled, but not treated | 3
Not completed — Dose data not recorded | 2

BASELINE CHARACTERISTICS:
Population: Analysis population included all treated participants.
Arm/Group | Mircera
Number analyzed (Participants) | 1285
Age, Continuous [Mean (Standard Deviation); unit: years] — Data for this baseline characteristic were available for 1276 participants only.
  years | 70.13 (13.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 570
  Male | 715

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Hemoglobin Cycling
Description: Hemoglobin cycling was defined as 1 or more cycles of oscillation in hemoglobin with an amplitude of greater than or equal to (>=) 1.5 gram per deciliter (g/dL) and a duration >=8 weeks.
Time Frame: 9 months
Population: Analysis population included all treated participants.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera
Number analyzed (Participants) | 1285
percentage of participants | 31.84

2. Secondary Outcome: Number of Full Hemoglobin Cycles Per Participant
Description: Hemoglobin cycling was defined as 1 or more cycles of oscillation in hemoglobin with an amplitude of >=1.5 g/dL and a duration >=8 weeks.
Time Frame: 9 months
Population: Analysis population included all treated participants.
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Mircera
Number analyzed (Participants) | 1285
cycles | 0.38 (0.61)

3. Secondary Outcome: Percentage of Participants With Type 2 Diabetes Who Experienced at Least 1 Hemoglobin Cycling
Description: as for outcome 2
Time Frame: 9 months
Population: Analysis population included all treated participants. 'N' (number of participants analyzed) included those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera
Number analyzed (Participants) | 207
percentage of participants | 29.83

ADVERSE EVENTS:
Description: Due to 'retrospective' nature of this registry data study, it was not possible to collect complete adverse events (AE) data. Hence, it was planned not to collect any AE data in this study.
Arm/Group | Mircera
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.